CLINICAL TRIAL: NCT02248831
Title: Non-invasive Evaluation of Cardiopulmonary Diseases Using Transthoracic Parametric Doppler Based Assessment of Lung Doppler Signals
Brief Title: Evaluation of Cardiopulmonary Diseases by Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Echosense Ltd. (Industry)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DOP19
Record Dates: First submitted 2014-09-18; First posted 2014-09-25 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2016-11

CONDITIONS: Dyspnea; Acute Decompensated Heart Failure
Keywords: Dyspnea; Acute decompensated heart failure; Doppler ultrasound; Lung Doppler signals
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Doppler ultrasound (Experimental): Using ultrasound noninvasively and recording Doppler signals from the right chest wall
  Interventions: Device: Recording Doppler ultrasound signals noninvasively

INTERVENTIONS:
Device: Recording Doppler ultrasound signals noninvasively — Using ultrasound noninvasively and recording Doppler signals from the right chest wall

SUMMARY:
Historically, ultrasound imaging of the lung parenchyma has been challenging because of the high total ultrasound energy attenuation and scattering by the air in the lungs. However, recent technological advancements have allowed for rapid assessment of various pulmonary diseases via the use of lung ultrasound. Furthermore, it has been shown that clear reproducible Doppler signals can be recorded from the lung parenchyma by means of a pulsed Doppler ultrasound system incorporating a special signal-processing package.

The LDS may contain information of significant diagnostic and physiological value regarding the pulmonary parenchyma and vasculature, as well as the cardio-vascular system in general. In a pilot clinical validation study of patients with acute decompensated heart failure (ADHF) patients, LDS signals unique to ADHF patients were identified, that superpose on the normal Lung Doppler Signals (unpublished data). These are high velocity "disorganized" variable signals that are not synchronous with the cardiac cycle but rather sometimes with respiration.

DETAILED DESCRIPTION:
Study Purpose and Rationale

The purpose of this study is to assess the utility of noninvasive assessment of lung Doppler signals performed via transthoracic parametric Doppler. The study has two major objectives and is thus, divided into two phases, which are on a continuum.

Phase 1: The objective is to further evaluate LDS among patients presenting to the emergency department with acute dyspnea, in order to determine the diagnostic value of this non-invasive method to distinguish cardiac from pulmonary causes of dyspnea.

Phase 2: In addition, for those patients admitted to the hospital with a clinical diagnosis of ADHF, we would like to further characterize changes in daily lung Doppler signal as a surrogate biomarker of intravascular volume status, as assessed by clinical assessment.

Study Design and Methods:

1. Overall study design

Phase 1:

Prospective cohort study of patients presenting to the Massachusetts General Hospital emergency department with acute dyspnea. . In addition, at MGH, pts admitted to the cardiac floors (Ellison 9, 10, 11) and general medicine floors (White 9, 10, 11) with an admitting diagnosis of heart failure, who presented with acute dyspnea, will be approached for enrollment within 24 hours of hospital admission. All patients with acute dyspnea will undergo routine clinical assessment, laboratory testing, and diagnostic imaging. In addition, all patients will also undergo transthoracic parametric Doppler ultrasound based assessment of LDS. Patients will be treated as usual, under the direction of the attending physician. Two independent cardiologists will perform detailed chart review on all patients to determine the etiology of acute dyspnea. They will be blinded to the results of the LDS. In the event of discrepant findings, a third cardiologist will perform a final detailed chart review to adjudicate the diagnosis.

Additionally, radiologist employed at MGH and who are independent to the study may perform blinded adjudication of the study participants' chest x-rays (CXR) obtained in the Emergency Department on the day of enrollment into the study

Phase 2:

In addition, patients diagnosed with ADHF (diagnosed based on the criteria described below), will undergo daily TPD and assessment of LDS to further characterize changes in LDS over time, until the day of discharge or up to day 7 of hospitalization, whichever comes first. In addition to the initial inpatient scans, study staff will try to acquire a final scan within 72 hours of discharge for patients diagnosed with ADHF, regardless of the day of hospitalization. This cohort of patients will also undergo daily clinical assessment of volume status, weight measurement, and BNP assessment. In the event that repeat BNP or NT-proBNP labs have not been drawn within 72 hours of discharge, study staff will coordinate with the pathology laboratory (Dr. Kent Lewandrowski) to perform the assay as a research test using excess clinical specimen from the subject's routine clinical blood draw if available. Research subjects will not be charged for the cost of the BNP or NT-Pro-BNP assay.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1(ED):

Inclusion criteria:

Age > 18 years Acute onset dyspnea

* Phase 2 (Inpatient):

Age > 18 years Acute onset dyspnea: defined as SOB at rest or with minimal activity, with onset within the past 14 days PLUS

The following criteria are required to be classified as heart failure (event has to meet all of the following criteria):

a) The patient exhibits documented new or worsening symptoms due to heart failure on presentation, including at least one of the following: i) Dyspnea (dyspnea with exertion, dyspnea at rest, orthopnea) ii) Decreased exercise tolerance b) The patient has objective evidence of new or worsening heart failure, consisting of at least two physical exam findings (or one physical exam finding and one diagnostic criterion) including: i) Physical exam findings considered to be due to heart failure, including new or worsened:

(1) Peripheral edema (2) Increasing abdominal distention or ascites (in the absence of primary hepatic disease) (3) Increased jugular venous pressure and/or hepatojugular reflux (4) Rapid weight gain thought to be related to fluid overload ii) Diagnostic findings considered to be due to heart failure, including new or worsened:

1. Increased B-type natriuretic peptide/ NT-proBNP concentrations consistent with decompensation of heart failure Note: In patients with chronically elevated natriuretic peptides, a significant increase should be noted above baseline.
2. Radiological evidence of pulmonary congestion

Exclusion Criteria:

* Phase 1 (ED):

Pregnant women Inability to consent

* Phase 2 (Inpatient):

Pregnant women Pneumonia - currently, or within the past 30 days Non-cardiogenic pulmonary edema (e.g. ARDS) Interstitial lung disease Inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2014-09; Primary Completion 2018-05 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Number of patients identified with COPD (or CHF) in comparison to physician diagnosis | 1y

SECONDARY OUTCOMES:
Identify changes in lung doppler signals according to the clinical status over few days in comparison to the physician diagnosis | 1y

CONTACTS AND LOCATIONS:
Overall Officials: Maulik Majmudar, Dr, Principal Investigator — MGH
Locations (1):
- Emergency Medicine department and Inpatients floors,MGH, Boston, Massachusetts, United States